CLINICAL TRIAL: NCT00606359
Title: Immunogenicity of the Inactivated Split-Virion Influenza Vaccine Administered by the Intradermal Route in Renal Transplant Subjects
Brief Title: Immunogenicity of the Inactivated Split-Virion Influenza Vaccine in Renal Transplant Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GID26
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Orthomyxoviridae Infections
Keywords: Influenza; Orthomyxoviridae Infections; Renal Transplant
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group 1 (Experimental)
  Interventions: Biological: Inactivated, split-virion influenza virus
- Study Group 2 (Active Comparator)
  Interventions: Biological: Inactivated, split-virion influenza virus

INTERVENTIONS:
Biological: Inactivated, split-virion influenza virus — 0.1 mL, Intradermal. 2 vaccinations 12 months apart
  Arms: Study Group 1
Biological: Inactivated, split-virion influenza virus — 0.5 mL, Intramuscular. 2 vaccinations, 12 months apart
  Other Names: Vaxigrip®
  Arms: Study Group 2

SUMMARY:
Primary Objective:

To describe the immunogenicity of an injection of the investigational inactivated, split-virion influenza vaccine 21 days after vaccination in 18 to 60 years old renal transplant subjects identified as non-responder to previous vaccination with the IM reference vaccine (Vaxigrip®).

Secondary Objective:

To describe the safety of an injection of the investigational inactivated, split-virion influenza vaccine in 18 to 60 years old renal transplant subjects identified as non-responder to previous vaccination with the IM reference vaccine

DETAILED DESCRIPTION:
The trial is a multicenter, randomized, controlled trial in renal transplant subjects aged 18 to 60 years who are non-responders to vaccination with the reference vaccine. Subjects will be randomized to receive either the 2007-2008 15 µg investigational vaccine or the 2007-2008 IM reference vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Able to attend all scheduled visits and to comply with all trial procedures.
* Subject with renal transplant for at least 6 months.
* Subject with stable renal function, i.e. with a variation of creatinin value < 20% and with a creatinin clearance estimated according to Cockroft and Gault calculation > 20 mL/min during the 3 months preceding inclusion.
* Aged 18 to 59 years on the day of the screening visit.
* Informed Consent Form signed.
* Subject entitled to national social security.
* Subject under immunosuppressive therapy.
* For a woman, inability to bear a child or negative urine pregnancy test.
* Subject non-responder to previous IM vaccination with the 2006-2007 Northern Hemisphere Vaxigrip® formulation.

Exclusion Criteria:

* Subject with sign of transplanted kidney reject within 3 months preceding vaccination according to medical practice.
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Febrile illness (oral temperature ≥ 37.5°C, or rectal equivalent temperature ≥ 38.0°C) on the day of inclusion.
* Breast-feeding.
* Participation in another clinical trial in the 4 weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Congenital immunodeficiency, anti-cancer chemotherapy or radiation therapy within the preceding 6 months.
* Chronic illness, except renal failure or renal disorders, at a stage that could interfere with trial conduct or completion.
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures.
* Blood or blood-derived products received in the past 3 months .
* Any vaccination in the 4 weeks preceding the trial vaccination.
* Vaccination planned in the 4 weeks following the trial vaccination.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular (IM) vaccination
* Previous vaccination against influenza in the preceding 6 months.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Anti-HA individual titers | 21 Days Post-vaccination 2
Individual titers ratio | 21 Days Post-vaccination 2
Seroconversion or significant increase | 21 Days Post-vaccination 2

SECONDARY OUTCOMES:
Safety: Adverse events in the first 21 days after each vaccination; Pre-listed reactions in the 7 days following each vaccination; Serious adverse events during the entire trial. | 21 days following each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Lyon, France

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com